CLINICAL TRIAL: NCT06034405
Title: Analysis of Lumbar Spine Stenosis Specimens for Identification of Transthyretin Cardiac Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mathew S. Maurer, MD, Arnold and Arlene Goldstein Professor of Cardiology (in Medicine, Dept of Medicine Cardiology), Columbia University
Other Study IDs: AAAU4704; R01AG081582-01 (NIH)
Record Dates: First submitted 2023-08-17; First posted 2023-09-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spinal Stenosis; Cardiac Amyloidosis; ATTR Amyloidosis Wild Type; ATTR Gene Mutation; ATTRV122I Amyloidosis; Cardiomyopathy, Hypertrophic
MeSH Terms: conditions — Spinal Stenosis; Amyloid Neuropathies, Familial; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn and analyzed for standard chemistry (Chem-7), liver function tests, NT-proBNP, troponin I and T, and TTR gene sequencing (see below). For subjects with ATTR-CA by positive uptake of 99mTc-PYP, further testing of prealbumin and monoclonal proteins (serum free light chains and immunofixation in serum and urine) will be performed. Additional aliquots will be stored at -80° for future analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATTR Negative: Participants who have undergone previous lumbar spinal, and/or carpel tunnel surgery will provide medical record data and spinal specimen for analysis of presence of ATTR amyloid.
- ATTR Positive: Participants who have undergone previous lumbar spinal, and/or carpel tunnel surgery will provide medical record data, spinal specimen, prospective data from cardiac workup with confirmed ATTR amyloid in spinal specimen then undergo cardiac workup for cardiac phenotyping/genotyping.
  Interventions: Diagnostic Test: Tc99-PYP or Tc99-HDMP Scan

INTERVENTIONS:
Diagnostic Test: Tc99-PYP or Tc99-HDMP Scan — Difference in ATTR-CA prevalence between subjects with TTR and indeterminate amyloid deposits in their spine by myocardial uptake of Tc99-PYP.
  Groups: ATTR Positive

SUMMARY:
Primary objective:

To identify older adults with transthyretin cardiac amyloidosis (ATTR-CA) early in the course of the illness, at a time when disease modifying therapies are most effective.

The specific aims of this epidemiologic investigation include:

1. To identify subjects with previous lumbar spinal stenosis (LSS) Surgery who have evidence of transthyretin (TTR) amyloid deposits in spinal specimens and could be at risk for ATTR cardiac amyloidosis.
2. To evaluate for ATTR-CA among those with localized TTR in the spinal tissue.

The study will also explore the following:

1. The prevalence of amyloid in lumbar spinal stenosis specimens by Congo Red staining.
2. The prevalence of TTR deposits among subjects with amyloid as determined by mass spectrometry.
3. Evaluation of a novel artificial intelligence technique for that can identify amyloid histologically with standard H&E staining.
4. Difference in ATTR-CA prevalence between subjects with TTR and indeterminate amyloid deposits in subject's spine by myocardial uptake of technetium pyrophosphate scan (Tc99-PYP).

DETAILED DESCRIPTION:
This is a multicenter, prospective cohort study aimed at facilitating identification of individuals with ATTR-CA. Investigators will identify subjects with previous LSS surgery who have evidence of TTR amyloid deposits in spinal specimens. Subjects with localized TTR in spinal tissue will be invited to an on-site visit and be evaluated for the presence of clinical manifestations of ATTR cardiac amyloidosis (ATTR-CA).

Subjects will undergo nuclear scintigraphy, TTR genetic test, a clinical evaluation, electrocardiogram, and echocardiogram. Quality of life questionnaires will also be administered. Subjects who have myocardial retention of the imaging radiotracer with a Perugini score equal to 2 (uptake equal to bone) or 3 (uptake greater than bone) and confirmation by SPECT or SPECT/CT that the uptake is myocardial in nature and have no evidence of monoclonal proteins will be diagnosed with ATTR-CA.

This study is to be conducted at five study sites: Boston Medical Center, Cedars Sinai Medical Center, Cleveland Clinic, Columbia University Irving Medical Center, and Tufts University Medical Center. The Mayo Clinic will serve a Pathology research core to analyze spine specimens.

Most of the subjects are expected to complete all the study procedures and questionnaires on a single day.

Up to 1663 patients will be consented in this study to have spinal specimens examined for the presence of amyloid by Congo Red at the Mayo Clinic core lab. From the pool of subjects with amyloid detected (which anticipate will be 33% or at least 544), the investigators expect to recruit 163 participants to undergo cardiac phenotyping (Tc99m and cardiac evaluation). Among the 163 participants who undergo cardiac phenotyping, 98 will have TTR as the precursor protein identified by mass spectrometry and 65 will have an indeterminant precursor protein by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically indicated spinal decompressive surgery within 20 years prior to enrollment.
2. Age ≥50 years at the time of the surgery.
3. Able to understand and sign the informed consent document after the nature of the study has been fully explained.

Exclusion Criteria:

The presence of any of the following excludes eligibility for enrollment in this study:

1. Confirmed primary amyloidosis (AL) or secondary amyloidosis (AA).
2. Known TTR amyloidosis.
3. Other reason that would make the subject inappropriate for entry into this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Previously procured surgical specimens from spinal surgery performed within 20 years prior to enrollment.
Sampling Method: Probability Sample
Enrollment: 1663 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects with previous LSS surgery who have evidence of TTR amyloid deposits in their spinal specimen and could be at risk for ATTR cardiac amyloidosis | up to 3 years
  To identify who can be at risk for ATTR Cardiac Amyloidosis. The investigator is going to collect spinal ligamentum flavum specimens and stain with congo red and those who result positive for ATTR amyloid in their spinal specimen will be counted

SECONDARY OUTCOMES:
Percent of subjects with ATTR-CA among those with localized TTR in their spinal tissue | up to 6 years
  To evaluate number of subjects with ATTR-CA among those with localized TTR in their spinal tissue. The investigator is going to perform standard of care (SOC) cardiac amyloidosis work up including PYP scan to confirm cardiac phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Mathew S Maurer, MD, Principal Investigator — Columbia University
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Upadhya B, Pisani B, Kitzman DW. Evolution of a Geriatric Syndrome: Pathophysiology and Treatment of Heart Failure with Preserved Ejection Fraction. J Am Geriatr Soc. 2017 Nov;65(11):2431-2440. doi: 10.1111/jgs.15141. PMID 29124734
- [Background] Ruberg FL, Grogan M, Hanna M, Kelly JW, Maurer MS. Transthyretin Amyloid Cardiomyopathy: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Jun 11;73(22):2872-2891. doi: 10.1016/j.jacc.2019.04.003. PMID 31171094
- [Background] Griffin JM, Rosenblum H, Maurer MS. Pathophysiology and Therapeutic Approaches to Cardiac Amyloidosis. Circ Res. 2021 May 14;128(10):1554-1575. doi: 10.1161/CIRCRESAHA.121.318187. Epub 2021 May 13. PMID 33983835
- [Background] AbouEzzeddine OF, Davies DR, Scott CG, Fayyaz AU, Askew JW, McKie PM, Noseworthy PA, Johnson GB, Dunlay SM, Borlaug BA, Chareonthaitawee P, Roger VL, Dispenzieri A, Grogan M, Redfield MM. Prevalence of Transthyretin Amyloid Cardiomyopathy in Heart Failure With Preserved Ejection Fraction. JAMA Cardiol. 2021 Nov 1;6(11):1267-1274. doi: 10.1001/jamacardio.2021.3070. PMID 34431962
- [Background] Gonzalez-Lopez E, Gallego-Delgado M, Guzzo-Merello G, de Haro-Del Moral FJ, Cobo-Marcos M, Robles C, Bornstein B, Salas C, Lara-Pezzi E, Alonso-Pulpon L, Garcia-Pavia P. Wild-type transthyretin amyloidosis as a cause of heart failure with preserved ejection fraction. Eur Heart J. 2015 Oct 7;36(38):2585-94. doi: 10.1093/eurheartj/ehv338. Epub 2015 Jul 28. PMID 26224076
- [Background] Castano A, Narotsky DL, Hamid N, Khalique OK, Morgenstern R, DeLuca A, Rubin J, Chiuzan C, Nazif T, Vahl T, George I, Kodali S, Leon MB, Hahn R, Bokhari S, Maurer MS. Unveiling transthyretin cardiac amyloidosis and its predictors among elderly patients with severe aortic stenosis undergoing transcatheter aortic valve replacement. Eur Heart J. 2017 Oct 7;38(38):2879-2887. doi: 10.1093/eurheartj/ehx350. PMID 29019612
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Griffin JM, Maurer MS. Transthyretin cardiac amyloidosis: A treatable form of heart failure with a preserved ejection fraction. Trends Cardiovasc Med. 2021 Jan;31(1):59-66. doi: 10.1016/j.tcm.2019.12.003. Epub 2019 Dec 17. PMID 31889610
- [Background] Adams D, Gonzalez-Duarte A, O'Riordan WD, Yang CC, Ueda M, Kristen AV, Tournev I, Schmidt HH, Coelho T, Berk JL, Lin KP, Vita G, Attarian S, Plante-Bordeneuve V, Mezei MM, Campistol JM, Buades J, Brannagan TH 3rd, Kim BJ, Oh J, Parman Y, Sekijima Y, Hawkins PN, Solomon SD, Polydefkis M, Dyck PJ, Gandhi PJ, Goyal S, Chen J, Strahs AL, Nochur SV, Sweetser MT, Garg PP, Vaishnaw AK, Gollob JA, Suhr OB. Patisiran, an RNAi Therapeutic, for Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):11-21. doi: 10.1056/NEJMoa1716153. PMID 29972753
- [Background] Benson MD, Waddington-Cruz M, Berk JL, Polydefkis M, Dyck PJ, Wang AK, Plante-Bordeneuve V, Barroso FA, Merlini G, Obici L, Scheinberg M, Brannagan TH 3rd, Litchy WJ, Whelan C, Drachman BM, Adams D, Heitner SB, Conceicao I, Schmidt HH, Vita G, Campistol JM, Gamez J, Gorevic PD, Gane E, Shah AM, Solomon SD, Monia BP, Hughes SG, Kwoh TJ, McEvoy BW, Jung SW, Baker BF, Ackermann EJ, Gertz MA, Coelho T. Inotersen Treatment for Patients with Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):22-31. doi: 10.1056/NEJMoa1716793. PMID 29972757
- [Background] Gillmore JD, Gane E, Taubel J, Kao J, Fontana M, Maitland ML, Seitzer J, O'Connell D, Walsh KR, Wood K, Phillips J, Xu Y, Amaral A, Boyd AP, Cehelsky JE, McKee MD, Schiermeier A, Harari O, Murphy A, Kyratsous CA, Zambrowicz B, Soltys R, Gutstein DE, Leonard J, Sepp-Lorenzino L, Lebwohl D. CRISPR-Cas9 In Vivo Gene Editing for Transthyretin Amyloidosis. N Engl J Med. 2021 Aug 5;385(6):493-502. doi: 10.1056/NEJMoa2107454. Epub 2021 Jun 26. PMID 34215024
- [Background] Maurer MS. Gene Editing - A Cure for Transthyretin Amyloidosis? N Engl J Med. 2021 Aug 5;385(6):558-559. doi: 10.1056/NEJMe2110557. No abstract available. PMID 34347958
- [Background] Maurer MS, Mann DL. The Tafamidis Drug Development Program: A Translational Triumph. JACC Basic Transl Sci. 2018 Dec 31;3(6):871-873. doi: 10.1016/j.jacbts.2018.10.001. eCollection 2018 Dec. No abstract available. PMID 30623146
- [Background] Nativi-Nicolau JN, Karam C, Khella S, Maurer MS. Screening for ATTR amyloidosis in the clinic: overlapping disorders, misdiagnosis, and multiorgan awareness. Heart Fail Rev. 2022 May;27(3):785-793. doi: 10.1007/s10741-021-10080-2. Epub 2021 Feb 20. PMID 33609196
- [Background] Donnelly JP, Hanna M, Sperry BW, Seitz WH Jr. Carpal Tunnel Syndrome: A Potential Early, Red-Flag Sign of Amyloidosis. J Hand Surg Am. 2019 Oct;44(10):868-876. doi: 10.1016/j.jhsa.2019.06.016. Epub 2019 Aug 7. PMID 31400950
- [Background] Sperry BW, Reyes BA, Ikram A, Donnelly JP, Phelan D, Jaber WA, Shapiro D, Evans PJ, Maschke S, Kilpatrick SE, Tan CD, Rodriguez ER, Monteiro C, Tang WHW, Kelly JW, Seitz WH Jr, Hanna M. Tenosynovial and Cardiac Amyloidosis in Patients Undergoing Carpal Tunnel Release. J Am Coll Cardiol. 2018 Oct 23;72(17):2040-2050. doi: 10.1016/j.jacc.2018.07.092. PMID 30336828
- [Background] Geller HI, Singh A, Alexander KM, Mirto TM, Falk RH. Association Between Ruptured Distal Biceps Tendon and Wild-Type Transthyretin Cardiac Amyloidosis. JAMA. 2017 Sep 12;318(10):962-963. doi: 10.1001/jama.2017.9236. PMID 28898370
- [Background] Rubin J, Alvarez J, Teruya S, Castano A, Lehman RA, Weidenbaum M, Geller JA, Helmke S, Maurer MS. Hip and knee arthroplasty are common among patients with transthyretin cardiac amyloidosis, occurring years before cardiac amyloid diagnosis: can we identify affected patients earlier? Amyloid. 2017 Dec;24(4):226-230. doi: 10.1080/13506129.2017.1375908. Epub 2017 Sep 14. PMID 28906148
- [Background] George KM, Dowd RS, Nail J, Yu A, Mastroianni M, Wang AY, Arkun K, Patel A, Kryzanski J, Comenzo R, Riesenburger RI. Wild-Type Transthyretin Amyloidosis Occurring in the Ligamentum Flavum of the Cervicothoracic Spine. World Neurosurg. 2020 Oct;142:e325-e330. doi: 10.1016/j.wneu.2020.06.228. Epub 2020 Jul 8. PMID 32652280
- [Background] George KM, Hernandez NS, Breton J, Cooper B, Dowd RS, Nail J, Yu A, Mastroianni M, Wang A, Godara A, Zhang D, Arkun K, Patel AR, Varga C, Soto O, Kryzanski J, Comenzo R, Riesenburger R. Lumbar ligamentum flavum burden: Evaluating the role of ATTRwt amyloid deposition in ligamentum flavum thickness at all lumbar levels. Clin Neurol Neurosurg. 2021 Jul;206:106708. doi: 10.1016/j.clineuro.2021.106708. Epub 2021 May 25. PMID 34053807
- [Background] Westermark P, Westermark GT, Suhr OB, Berg S. Transthyretin-derived amyloidosis: probably a common cause of lumbar spinal stenosis. Ups J Med Sci. 2014 Aug;119(3):223-8. doi: 10.3109/03009734.2014.895786. Epub 2014 Mar 12. PMID 24620715
- [Background] Yanagisawa A, Ueda M, Sueyoshi T, Okada T, Fujimoto T, Ogi Y, Kitagawa K, Tasaki M, Misumi Y, Oshima T, Jono H, Obayashi K, Hirakawa K, Uchida H, Westermark P, Ando Y, Mizuta H. Amyloid deposits derived from transthyretin in the ligamentum flavum as related to lumbar spinal canal stenosis. Mod Pathol. 2015 Feb;28(2):201-7. doi: 10.1038/modpathol.2014.102. Epub 2014 Sep 5. PMID 25189643
- [Background] Basdavanos A, Maurer MS, Ives L, Derwin K, Ricchetti ET, Seitz W, Hanna M. Prevalence of Orthopedic Manifestations in Patients With Cardiac Amyloidosis With a Focus on Shoulder Pathologies. Am J Cardiol. 2023 Mar 1;190:67-74. doi: 10.1016/j.amjcard.2022.11.014. Epub 2022 Dec 23. PMID 36566619
- [Background] Westin O, Fosbol EL, Maurer MS, Leicht BP, Hasbak P, Mylin AK, Rorvig S, Lindkaer TH, Johannesen HH, Gustafsson F. Screening for Cardiac Amyloidosis 5 to 15 Years After Surgery for Bilateral Carpal Tunnel Syndrome. J Am Coll Cardiol. 2022 Sep 6;80(10):967-977. doi: 10.1016/j.jacc.2022.06.026. PMID 36049804
- [Background] Bhuiyan T, Helmke S, Patel AR, Ruberg FL, Packman J, Cheung K, Grogan D, Maurer MS. Pressure-volume relationships in patients with transthyretin (ATTR) cardiac amyloidosis secondary to V122I mutations and wild-type transthyretin: Transthyretin Cardiac Amyloid Study (TRACS). Circ Heart Fail. 2011 Mar;4(2):121-8. doi: 10.1161/CIRCHEARTFAILURE.109.910455. Epub 2010 Dec 29. PMID 21191093
- [Background] Hilmy AM, el-Domiaty NA, Daabees AY, Abou Taleb EM. The use of the chelating agent EDTA in the treatment of acute cadmium toxicity, tissue distribution and some blood parameters in the Egyptian toad Bufo regularis. Comp Biochem Physiol C Comp Pharmacol Toxicol. 1986;85(1):67-74. doi: 10.1016/0742-8413(86)90053-8. PMID 2877808
- [Background] Saith SE, Maurer MS, Patel AR. Systemic Amyloidosis due to Monoclonal Immunoglobulins: Cardiac Involvement. Hematol Oncol Clin North Am. 2020 Dec;34(6):1055-1068. doi: 10.1016/j.hoc.2020.07.006. Epub 2020 Sep 14. PMID 33099423
- [Background] Hanna M, Damy T, Grogan M, Stewart M, Gundapaneni B, Patterson TA, Schwartz JH, Sultan MB, Maurer MS. Impact of Tafamidis on Health-Related Quality of Life in Patients With Transthyretin Amyloid Cardiomyopathy (from the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial). Am J Cardiol. 2021 Feb 15;141:98-105. doi: 10.1016/j.amjcard.2020.10.066. Epub 2020 Nov 19. PMID 33220323
- [Background] Hanna M, Damy T, Grogan M, Stewart M, Gundapaneni B, Sultan MB, Maurer MS. Tafamidis and quality of life in people with transthyretin amyloid cardiomyopathy in the study ATTR-ACT: A plain language summary. Future Cardiol. 2022 Mar;18(3):165-172. doi: 10.2217/fca-2021-0095. Epub 2021 Nov 15. PMID 34779246
- [Background] Hanna M, Ruberg FL, Maurer MS, Dispenzieri A, Dorbala S, Falk RH, Hoffman J, Jaber W, Soman P, Witteles RM, Grogan M. Cardiac Scintigraphy With Technetium-99m-Labeled Bone-Seeking Tracers for Suspected Amyloidosis: JACC Review Topic of the Week. J Am Coll Cardiol. 2020 Jun 9;75(22):2851-2862. doi: 10.1016/j.jacc.2020.04.022. PMID 32498813
- [Background] Hartnett J, Jaber W, Maurer M, Sperry B, Hanna M, Collier P, Patel DR, Wazni OM, Donnellan E. Electrophysiological Manifestations of Cardiac Amyloidosis: JACC: CardioOncology State-of-the-Art Review. JACC CardioOncol. 2021 Oct 19;3(4):506-515. doi: 10.1016/j.jaccao.2021.07.010. eCollection 2021 Oct. PMID 34729522
- [Background] Judge DP, Heitner SB, Falk RH, Maurer MS, Shah SJ, Witteles RM, Grogan M, Selby VN, Jacoby D, Hanna M, Nativi-Nicolau J, Patel J, Rao S, Sinha U, Turtle CW, Fox JC. Transthyretin Stabilization by AG10 in Symptomatic Transthyretin Amyloid Cardiomyopathy. J Am Coll Cardiol. 2019 Jul 23;74(3):285-295. doi: 10.1016/j.jacc.2019.03.012. Epub 2019 Mar 15. PMID 30885685
- [Background] Judge DP, Kristen AV, Grogan M, Maurer MS, Falk RH, Hanna M, Gillmore J, Garg P, Vaishnaw AK, Harrop J, Powell C, Karsten V, Zhang X, Sweetser MT, Vest J, Hawkins PN. Phase 3 Multicenter Study of Revusiran in Patients with Hereditary Transthyretin-Mediated (hATTR) Amyloidosis with Cardiomyopathy (ENDEAVOUR). Cardiovasc Drugs Ther. 2020 Jun;34(3):357-370. doi: 10.1007/s10557-019-06919-4. PMID 32062791
- [Background] Maurer MS, Hanna M, Grogan M, Dispenzieri A, Witteles R, Drachman B, Judge DP, Lenihan DJ, Gottlieb SS, Shah SJ, Steidley DE, Ventura H, Murali S, Silver MA, Jacoby D, Fedson S, Hummel SL, Kristen AV, Damy T, Plante-Bordeneuve V, Coelho T, Mundayat R, Suhr OB, Waddington Cruz M, Rapezzi C; THAOS Investigators. Genotype and Phenotype of Transthyretin Cardiac Amyloidosis: THAOS (Transthyretin Amyloid Outcome Survey). J Am Coll Cardiol. 2016 Jul 12;68(2):161-72. doi: 10.1016/j.jacc.2016.03.596. PMID 27386769
- [Background] Sueyoshi T, Ueda M, Jono H, Irie H, Sei A, Ide J, Ando Y, Mizuta H. Wild-type transthyretin-derived amyloidosis in various ligaments and tendons. Hum Pathol. 2011 Sep;42(9):1259-64. doi: 10.1016/j.humpath.2010.11.017. Epub 2011 Feb 21. PMID 21334722
- [Background] Garcia-Pavia P, Rapezzi C, Adler Y, Arad M, Basso C, Brucato A, Burazor I, Caforio ALP, Damy T, Eriksson U, Fontana M, Gillmore JD, Gonzalez-Lopez E, Grogan M, Heymans S, Imazio M, Kindermann I, Kristen AV, Maurer MS, Merlini G, Pantazis A, Pankuweit S, Rigopoulos AG, Linhart A. Diagnosis and treatment of cardiac amyloidosis. A position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur J Heart Fail. 2021 Apr;23(4):512-526. doi: 10.1002/ejhf.2140. Epub 2021 Apr 7. PMID 33826207
- [Background] Kittleson MM, Maurer MS, Ambardekar AV, Bullock-Palmer RP, Chang PP, Eisen HJ, Nair AP, Nativi-Nicolau J, Ruberg FL; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology. Cardiac Amyloidosis: Evolving Diagnosis and Management: A Scientific Statement From the American Heart Association. Circulation. 2020 Jul 7;142(1):e7-e22. doi: 10.1161/CIR.0000000000000792. Epub 2020 Jun 1. PMID 32476490
- [Background] Rapezzi C, Aimo A, Serenelli M, Barison A, Vergaro G, Passino C, Panichella G, Sinagra G, Merlo M, Fontana M, Gillmore J, Quarta CC, Maurer MS, Kittleson MM, Garcia-Pavia P, Emdin M. Critical Comparison of Documents From Scientific Societies on Cardiac Amyloidosis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Apr 5;79(13):1288-1303. doi: 10.1016/j.jacc.2022.01.036. PMID 35361352
- [Background] Nativi-Nicolau J, Siu A, Dispenzieri A, Maurer MS, Rapezzi C, Kristen AV, Garcia-Pavia P, LoRusso S, Waddington-Cruz M, Lairez O, Witteles R, Chapman D, Amass L, Grogan M; THAOS Investigators. Temporal Trends of Wild-Type Transthyretin Amyloid Cardiomyopathy in the Transthyretin Amyloidosis Outcomes Survey. JACC CardioOncol. 2021 Oct 19;3(4):537-546. doi: 10.1016/j.jaccao.2021.08.009. eCollection 2021 Oct. PMID 34729526
- [Background] Maurer MS, Elliott P, Comenzo R, Semigran M, Rapezzi C. Addressing Common Questions Encountered in the Diagnosis and Management of Cardiac Amyloidosis. Circulation. 2017 Apr 4;135(14):1357-1377. doi: 10.1161/CIRCULATIONAHA.116.024438. PMID 28373528
- [Background] Lane T, Fontana M, Martinez-Naharro A, Quarta CC, Whelan CJ, Petrie A, Rowczenio DM, Gilbertson JA, Hutt DF, Rezk T, Strehina SG, Caringal-Galima J, Manwani R, Sharpley FA, Wechalekar AD, Lachmann HJ, Mahmood S, Sachchithanantham S, Drage EPS, Jenner HD, McDonald R, Bertolli O, Calleja A, Hawkins PN, Gillmore JD. Natural History, Quality of Life, and Outcome in Cardiac Transthyretin Amyloidosis. Circulation. 2019 Jul 2;140(1):16-26. doi: 10.1161/CIRCULATIONAHA.118.038169. Epub 2019 May 21. PMID 31109193
- [Background] Rubin J, Maurer MS. Cardiac Amyloidosis: Overlooked, Underappreciated, and Treatable. Annu Rev Med. 2020 Jan 27;71:203-219. doi: 10.1146/annurev-med-052918-020140. PMID 31986086
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Vrana JA, Gamez JD, Madden BJ, Theis JD, Bergen HR 3rd, Dogan A. Classification of amyloidosis by laser microdissection and mass spectrometry-based proteomic analysis in clinical biopsy specimens. Blood. 2009 Dec 3;114(24):4957-9. doi: 10.1182/blood-2009-07-230722. Epub 2009 Oct 1. PMID 19797517
- [Background] Campanella G, Hanna MG, Geneslaw L, Miraflor A, Werneck Krauss Silva V, Busam KJ, Brogi E, Reuter VE, Klimstra DS, Fuchs TJ. Clinical-grade computational pathology using weakly supervised deep learning on whole slide images. Nat Med. 2019 Aug;25(8):1301-1309. doi: 10.1038/s41591-019-0508-1. Epub 2019 Jul 15. PMID 31308507
- [Background] Miller AB, Januzzi JL, O'Neill BJ, Gundapaneni B, Patterson TA, Sultan MB, Lopez-Sendon J. Causes of Cardiovascular Hospitalization and Death in Patients With Transthyretin Amyloid Cardiomyopathy (from the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial [ATTR-ACT]). Am J Cardiol. 2021 Jun 1;148:146-150. doi: 10.1016/j.amjcard.2021.02.035. Epub 2021 Mar 3. PMID 33667442
- [Background] Kubo SH, Schulman S, Starling RC, Jessup M, Wentworth D, Burkhoff D. Development and validation of a patient questionnaire to determine New York Heart Association classification. J Card Fail. 2004 Jun;10(3):228-35. doi: 10.1016/j.cardfail.2003.10.005. PMID 15190533
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Carroll JD, Gaasch WH, McAdam KP. Amyloid cardiomyopathy: characterization by a distinctive voltage/mass relation. Am J Cardiol. 1982 Jan;49(1):9-13. doi: 10.1016/0002-9149(82)90270-3. PMID 6459025
- [Background] Amundsen BH, Helle-Valle T, Edvardsen T, Torp H, Crosby J, Lyseggen E, Stoylen A, Ihlen H, Lima JA, Smiseth OA, Slordahl SA. Noninvasive myocardial strain measurement by speckle tracking echocardiography: validation against sonomicrometry and tagged magnetic resonance imaging. J Am Coll Cardiol. 2006 Feb 21;47(4):789-93. doi: 10.1016/j.jacc.2005.10.040. Epub 2006 Jan 26. PMID 16487846
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077
- [Background] Devereux RB, Alonso DR, Lutas EM, Gottlieb GJ, Campo E, Sachs I, Reichek N. Echocardiographic assessment of left ventricular hypertrophy: comparison to necropsy findings. Am J Cardiol. 1986 Feb 15;57(6):450-8. doi: 10.1016/0002-9149(86)90771-x. PMID 2936235
- [Background] Mor-Avi V, Sugeng L, Weinert L, MacEneaney P, Caiani EG, Koch R, Salgo IS, Lang RM. Fast measurement of left ventricular mass with real-time three-dimensional echocardiography: comparison with magnetic resonance imaging. Circulation. 2004 Sep 28;110(13):1814-8. doi: 10.1161/01.CIR.0000142670.65971.5F. Epub 2004 Sep 20. PMID 15381653
- [Background] Takeuchi M, Nishikage T, Mor-Avi V, Sugeng L, Weinert L, Nakai H, Salgo IS, Gerard O, Lang RM. Measurement of left ventricular mass by real-time three-dimensional echocardiography: validation against magnetic resonance and comparison with two-dimensional and m-mode measurements. J Am Soc Echocardiogr. 2008 Sep;21(9):1001-5. doi: 10.1016/j.echo.2008.07.008. PMID 18765176
- [Background] Tendler A, Helmke S, Teruya S, Alvarez J, Maurer MS. The myocardial contraction fraction is superior to ejection fraction in predicting survival in patients with AL cardiac amyloidosis. Amyloid. 2015 Mar;22(1):61-6. doi: 10.3109/13506129.2014.994202. Epub 2014 Dec 16. PMID 25510353
- [Background] Bokhari S, Castano A, Pozniakoff T, Deslisle S, Latif F, Maurer MS. (99m)Tc-pyrophosphate scintigraphy for differentiating light-chain cardiac amyloidosis from the transthyretin-related familial and senile cardiac amyloidoses. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):195-201. doi: 10.1161/CIRCIMAGING.112.000132. Epub 2013 Feb 11. PMID 23400849
- [Background] Cheng RK, Levy WC, Vasbinder A, Teruya S, De Los Santos J, Leedy D, Maurer MS. Diuretic Dose and NYHA Functional Class Are Independent Predictors of Mortality in Patients With Transthyretin Cardiac Amyloidosis. JACC CardioOncol. 2020 Sep;2(3):414-424. doi: 10.1016/j.jaccao.2020.06.007. Epub 2020 Sep 15. PMID 33073249
- [Background] Lee JY, Moon SH, Suh BK, Yang MH, Park MS. Outcome and Complications in Surgical Treatment of Lumbar Stenosis or Spondylolisthesis in Geriatric Patients. Yonsei Med J. 2015 Sep;56(5):1199-205. doi: 10.3349/ymj.2015.56.5.1199. PMID 26256960
- [Background] Kazi DS, Bellows BK, Baron SJ, Shen C, Cohen DJ, Spertus JA, Yeh RW, Arnold SV, Sperry BW, Maurer MS, Shah SJ. Cost-Effectiveness of Tafamidis Therapy for Transthyretin Amyloid Cardiomyopathy. Circulation. 2020 Apr 14;141(15):1214-1224. doi: 10.1161/CIRCULATIONAHA.119.045093. Epub 2020 Feb 12. PMID 32078382
- [Background] Ruiz-Negron N, Nativi-Nicolau J, Maurer MS, Moran AE, Kovacsovics T, Bellows BK. Cost-effectiveness of technetium pyrophosphate scintigraphy versus heart biopsy for the diagnosis of transthyretin amyloidosis. Amyloid. 2019;26(sup1):71-72. doi: 10.1080/13506129.2019.1583192. No abstract available. PMID 31343305
- [Background] Weintraub WS, Bhatt DL, Zhang Z, Dolman S, Boden WE, Bress AP, King JB, Bellows BK, Tajeu GS, Derington CG, Johnson J, Andrade K, Steg PG, Miller M, Brinton EA, Jacobson TA, Tardif JC, Ballantyne CM, Kolm P. Cost-effectiveness of Icosapent Ethyl for High-risk Patients With Hypertriglyceridemia Despite Statin Treatment. JAMA Netw Open. 2022 Feb 1;5(2):e2148172. doi: 10.1001/jamanetworkopen.2021.48172. PMID 35157055
- [Background] Zhang Z, Kolm P, Grau-Sepulveda MV, Ponirakis A, O'Brien SM, Klein LW, Shaw RE, McKay C, Shahian DM, Grover FL, Mayer JE, Garratt KN, Hlatky M, Edwards FH, Weintraub WS. Cost-effectiveness of revascularization strategies: the ASCERT study. J Am Coll Cardiol. 2015 Jan 6;65(1):1-11. doi: 10.1016/j.jacc.2014.09.078. PMID 25572503
- [Background] Zhang Z, Kolm P, Boden WE, Hartigan PM, Maron DJ, Spertus JA, O'Rourke RA, Shaw LJ, Sedlis SP, Mancini GB, Berman DS, Dada M, Teo KK, Weintraub WS. The cost-effectiveness of percutaneous coronary intervention as a function of angina severity in patients with stable angina. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):172-82. doi: 10.1161/CIRCOUTCOMES.110.940502. Epub 2011 Feb 8. PMID 21304091